CLINICAL TRIAL: NCT03279978
Title: Phase Ib Evaluation of the Safety and Tolerability and Effect on Midazolam Metabolism of the Administration of Multiple Rising Doses of BI 730357 to Healthy Volunteers
Brief Title: This Study Tests How Healthy Men Tolerate Different Doses of BI 730357 and How the Metabolism of Midazolam is Affected by BI 730357
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1407-0002; 2017-001653-14 (EudraCT Number)
Record Dates: First submitted 2017-09-11; First posted 2017-09-12 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- BI 730357 25 mg fast (Experimental): Subjects were orally administered BI 730357 25 mg, film-coated tablet once daily over 14 days after a fasting period of at least 6 hours
  Interventions: Drug: BI 730357
- Placebo fast (Placebo Comparator): Subjects were orally administered matching Placebo to BI 730357, film-coated tablet after a fasting period of at least 6 hours.
  Interventions: Drug: Placebo
- Placebo fed (Placebo Comparator): Subjects were orally administered matching Placebo to BI 730357, film-coated tablet after the intake of a standard continental breakfast.
  Interventions: Drug: Placebo
- BI 730357 50 mg fast (Experimental): Subjects were orally administered BI 730357 50 mg, film-coated tablet once daily over 14 days after a fasting period of at least 6 hours.
  Interventions: Drug: BI 730357
- BI 730357 50mg/Placebo (Experimental): Subject was orally administered mixed treatment of BI 730357 50 mg and placebo, film-coated tablet once daily over 14 days after a fasting period of at least 6 hours
  Interventions: Drug: BI 730357; Drug: Placebo
- BI 730357 50 mg fed (Experimental): Subjects were orally administered BI 730357 50 mg, film-coated tablet once daily over 14 days after the intake of a standard continental breakfast.
  Interventions: Drug: BI 730357
- BI 730357 100 mg fast (Experimental): Subjects were orally administered BI 730357 100 mg, film-coated tablet once daily over 14 days after a fasting period of at least 6 hours
  Interventions: Drug: BI 730357
- BI 730357 200 mg fast (Experimental): Subjects were orally administered BI 730357 200 mg, film-coated tablet once daily over 28 days after a fasting period of at least 6 hours
  Interventions: Drug: BI 730357
- BI 730357 200 mg fed (Experimental): Subjects were orally administered a microdose of midazolam 75 microgram (75 μg) solution for injection, orally on Day -1, and prior receiving BI 730357 on Days 3, and 14. Subjects were orally administered BI 730357 200 mg, film-coated tablet once daily over 28 days after the intake of a standard continental breakfast.
  Interventions: Drug: BI 730357; Drug: Midazolam
- BI 730357 400 mg fed (Experimental): Subjects were orally administered a microdose of midazolam 75 microgram (75 μg) solution for injection, orally on Day -1, and prior receiving BI 730357 on Days 3, and 14. Subjects were orally administered BI 730357 400 mg, film-coated tablet once daily over 28 days after the intake of a standard continental breakfast.
  Interventions: Drug: BI 730357; Drug: Midazolam

INTERVENTIONS:
Drug: BI 730357 — BI 730357 film-coated tablet
  Arms: BI 730357 100 mg fast; BI 730357 200 mg fast; BI 730357 200 mg fed; BI 730357 25 mg fast; BI 730357 400 mg fed; BI 730357 50 mg fast; BI 730357 50 mg fed; BI 730357 50mg/Placebo
Drug: Placebo — Placebo
  Arms: BI 730357 50mg/Placebo; Placebo fast; Placebo fed
Drug: Midazolam — Once per day (QD) on Days -1, 3, and 14. Dose groups BI 730357 200 mg fed and BI 730357 400 mg fed
  Arms: BI 730357 200 mg fed; BI 730357 400 mg fed

SUMMARY:
Phase Ib evaluation of the safety, tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) properties of Multiple Rising Dose (MRD) administration of BI 730357 to healthy volunteers for up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the Investigator, based on a complete medical history, physical examination, vital signs (blood pressure, pulse rate), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Subjects with a partner who is a woman of childbearing potential (WOCBP) must be willing to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication
* Age of 18 to 45 years (incl.) at screening
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.) at screening
* Signed and dated written informed consent prior to admission to the study in accordance with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation

Exclusion criteria

* Any finding in the medical examination (including blood pressure, pulse rate or Electrocardiogram (ECG)) deviating from normal and judged as clinically relevant by the Investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the Investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the Investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract (except appendectomy and simple hernia repair) that could interfere with the PK of the trial medication
* Diseases of the Central Nervous System (CNS) (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or acute infections which are of relevance in the opinion of the Investigator
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc (corrected QT interval) interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Tobacco usage (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the Investigator; for instance, is considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Unwillingness to adhere to the rules of UV-light protection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CTC North GmbH & Co. KG, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Ooi QX, Kristoffersson A, Korell J, Flack M, L Plan E, Weber B. Bounded integer model-based analysis of psoriasis area and severity index in patients with moderate-to-severe plaque psoriasis receiving BI 730357. CPT Pharmacometrics Syst Pharmacol. 2023 Jun;12(6):758-769. doi: 10.1002/psp4.12948. Epub 2023 May 1. PMID 36919398
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, placebo-controlled, double-blind design investigating multiple rising doses
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist site to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Period: Overall Study
Arm/Group | Placebo Fast | Placebo Fed | BI 730357 25 mg Fast | BI 730357 50 mg Fast | BI 730357 50mg/Placebo | BI 730357 50 mg Fed | BI 730357 100 mg Fast | BI 730357 200 mg Fast | BI 730357 200 mg Fed | BI 730357 400 mg Fed
Started | 11 | 9 | 9 | 9 | 1 | 8 | 9 | 9 | 9 | 9
Completed | 10 | 8 | 8 | 9 | 1 | 8 | 8 | 9 | 9 | 8
Not Completed | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other than stated above | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Fast | Placebo Fed | BI 730357 25 mg Fast | BI 730357 50 mg Fast | BI 730357 50mg/Placebo | BI 730357 50 mg Fed | BI 730357 100 mg Fast | BI 730357 200 mg Fast | BI 730357 200 mg Fed | BI 730357 400 mg Fed | Total
Number analyzed (Participants) | 11 | 9 | 9 | 9 | 1 | 8 | 9 | 9 | 9 | 9 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.8 (7.6) | 26.8 (5.4) | 33.3 (7.0) | 32.3 (7.7) | 25.0 (NA) — only one patient received mixed treatment thus Standard deviation is not calculable | 25.4 (3.6) | 27.3 (2.2) | 27.1 (5.9) | 25.6 (4.4) | 30.6 (8.5) | 29.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 11 | 9 | 9 | 9 | 1 | 8 | 9 | 9 | 9 | 9 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 9 | 9 | 8 | 1 | 8 | 9 | 9 | 9 | 9 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4
  White | 10 | 7 | 9 | 8 | 1 | 7 | 8 | 8 | 7 | 9 | 74
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug-related Adverse Events (AEs)
Description: Number of subjects with drug-related Adverse Events (AEs) assessed by the investigator.
Time Frame: From first drug administration until 7 days after last dose, up to 21 days (for 25, 50 and 100 mg dose groups) and up to 35 days (for 200 and 400 mg dose groups)
Population: Treated Set: This subject set included all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment. (One subject was orally administered mixed treatment of BI 730357 50 mg fast and placebo fast, thus evaluated twice in each respective treatment arm)
Measure: Number; unit: Participants
Arm/Group | Placebo Fast | Placebo Fed | BI 730357 25 mg Fast | BI 730357 50 mg Fast | BI 730357 50 mg Fed | BI 730357 100 mg Fast | BI 730357 200 mg Fast | BI 730357 200 mg Fed | BI 730357 400 mg Fed
Number analyzed (Participants) | 12 | 9 | 9 | 10 | 8 | 9 | 9 | 9 | 9
Participants | 4 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 2

2. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte BI 730357 in Plasma Over a Uniform Dosing Interval Tau After Administration of the First Dose (AUCtau,1)
Description: Area under the concentration-time curve of the analyte BI 730357 in plasma over a uniform dosing interval tau after administration of the first dose (AUCtau,1).
  In this study AUCtau,1 = AUC0-24
Time Frame: -0.5h before dosing and 0.25h, 0.5h, 1h, 1.5h, 2 h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h and 23.5h after first dosing on Day1.
Population: Pharmacokinetic analysis set (PKS): all subjects from the treated set (TS) who provided at least one evaluable secondary pharmacokinetic endpoint and did not have an important protocol deviation relevant for the evaluation of pharmacokinetics. Arm: BI 730357 50mg/Placebo: This arm comprised 1 subject that was excluded from the PKS due the important protocol deviation of having received a mixed treatment (placebo and investigational drug), therefore was not included in the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole (nmol)·hour (h)/ liter(L)
Arm/Group | BI 730357 25 mg Fast | BI 730357 50 mg Fast | BI 730357 50 mg Fed | BI 730357 100 mg Fast | BI 730357 200 mg Fast | BI 730357 200 mg Fed | BI 730357 400 mg Fed
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 9 | 9 | 9
Nanomole (nmol)·hour (h)/ liter(L) | 2150 (31.2) | 3590 (34.4) | 4620 (27.9) | 6650 (26.4) | 9240 (32.2) | 11900 (22.6) | 15600 (24.5)
Statistical Analysis 1: Comparison: BI 730357 25 mg Fast vs BI 730357 50 mg Fast vs BI 730357 100 mg Fast vs BI 730357 200 mg Fast; Dose proportionality for AUC0-24 of BI 730357 in plasma - fasted groups was assessed using a power model (regression model applied to log-transformed data). In this study AUCtau,1 = AUC0-24; Test type: Other; Slope = 0.7124, 95% CI 2-sided [0.5702 to 0.8546], Standard Error of Mean 0.0694; Standard error of the mean is actually standard error of the slope. Based on the estimate for the slope parameter, a two sided 95% confidence interval for the slope was computed. Perfect dose proportionality would correspond to a slope of 1
Statistical Analysis 2: Comparison: BI 730357 50 mg Fed vs BI 730357 200 mg Fed vs BI 730357 400 mg Fed; Dose proportionality for AUC0-24 of BI 730357 in plasma - fed groups was assessed using a power model (regression model applied to log-transformed data). In this study AUCtau,1 = AUC0-24; Test type: Other; Slope = 0.5964, 95% CI 2-sided [0.4777 to 0.7151], Standard Error of Mean 0.0575; [other analysis details as in outcome 2, analysis 1]

3. Secondary Outcome: Maximum Measured Concentration of the Analyte BI 730357 in Plasma After Administration of the First Dose (Cmax)
Description: Maximum measured concentration of the analyte BI 730357 in plasma after administration of the first dose (Cmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole (nmol)/liter(L)
Arm/Group | BI 730357 25 mg Fast | BI 730357 50 mg Fast | BI 730357 50 mg Fed | BI 730357 100 mg Fast | BI 730357 200 mg Fast | BI 730357 200 mg Fed | BI 730357 400 mg Fed
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 9 | 9 | 9
Nanomole (nmol)/liter(L) | 143 (25.4) | 247 (37.6) | 368 (34.8) | 408 (32.5) | 537 (26.8) | 953 (36.5) | 1320 (24.0)
Statistical Analysis 1: Comparison: BI 730357 25 mg Fast vs BI 730357 50 mg Fast vs BI 730357 100 mg Fast vs BI 730357 200 mg Fast; Dose proportionality for Cmax of BI 730357 in plasma - fasted groups was assessed using a power model (regression model applied to log-transformed data); Test type: Other; Slope = 0.6445, 95% CI 2-sided [0.5124 to 0.7766], Standard Error of Mean 0.0649; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 730357 50 mg Fed vs BI 730357 200 mg Fed vs BI 730357 400 mg Fed; Dose proportionality for Cmax of BI 730357 in plasma - fed groups was assessed using a power model (regression model applied to log-transformed data); Test type: Other; Slope = 0.6223, 95% CI 2-sided [0.4747 to 0.7699], Standard Error of Mean 0.0715; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 730357 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss) After Last Dose Administration.
Description: Area under the concentration-time curve of BI 730357 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) after last dose administration is reported. τ for 25, 50, 100 , 200 and 400 mg dose groups is: 24 hours (h).
  Time Frame: For 25, 50, and 100 mg dose groups: -0.5h before dosing and 0.25h, 0.5h, 1h, 1.5h, 2 h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 23.5h, 47.5 and 71.5 h after last dose on Day14. For 200 and 400 mg dose groups: -0.5h before last dose and 1.0h, 2.0h, 3.0h, 4.0h and 24.0h after last dose on Day28.
Time Frame: Day 14 and Day 28 (Please refer description for the time frame in detail)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole (nmol)·hour (h)/ liter(L)
Arm/Group | BI 730357 25 mg Fast | BI 730357 50 mg Fast | BI 730357 50 mg Fed | BI 730357 100 mg Fast | BI 730357 200 mg Fast | BI 730357 200 mg Fed | BI 730357 400 mg Fed
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 7 | 8 | 9
Nanomole (nmol)·hour (h)/ liter(L) | 4200 (50.0) | 7550 (30.3) | 9950 (29.4) | 14100 (24.5) | 14600 (45.0) | 29700 (30.0) | 31400 (38.2)
Statistical Analysis 1: Comparison: BI 730357 25 mg Fast vs BI 730357 50 mg Fast vs BI 730357 100 mg Fast vs BI 730357 200 mg Fast; Dose proportionality for AUCτ,ss of BI 730357 in plasma - fasted groups was assessed using a power model (regression model applied to log-transformed data); Test type: Other; Slope = 0.6401, 95% CI 2-sided [0.4545 to 0.8258], Standard Error of Mean 0.0909; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 730357 50 mg Fed vs BI 730357 200 mg Fed vs BI 730357 400 mg Fed; Dose proportionality for AUCτ,ss of BI 730357 in plasma - fed groups was assessed using a power model (regression model applied to log-transformed data); Test type: Other; Slope = 0.5811, 95% CI 2-sided [0.4013 to 0.7609], Standard Error of Mean 0.0864; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: Maximum Measured Concentration of the Analyte BI 730357 in Plasma at Steady State Over a Uniform Dosing Interval τ After the Last Dose (Cmax,ss)
Description: Maximum measured concentration of BI 730357 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) after last dose administration is reported. τ for 25, 50, 100 , 200 and 400 mg dose groups is: 24 hours (h).
  Time Frame:
  For 25, 50, and 100 mg dose groups:-0.5h before dosing and 0.25h, 0.5h, 1h, 1.5h, 2 h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 12h, 23.5h, 47.5 and 71.5 h after last dose on Day14.
  For 200 and 400 mg dose groups: -0.5h before last dose and 1.0h, 2.0h, 3.0h, 4.0h and 24.0h after last dose on Day28.
Time Frame: Day 14 and Day 28 (Please refer description for the time frame in detail)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole (nmol)/ liter(L)
Arm/Group | BI 730357 25 mg Fast | BI 730357 50 mg Fast | BI 730357 50 mg Fed | BI 730357 100 mg Fast | BI 730357 200 mg Fast | BI 730357 200 mg Fed | BI 730357 400 mg Fed
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 9 | 9 | 9
Nanomole (nmol)/ liter(L) | 277 (37.6) | 474 (26.7) | 697 (26.5) | 793 (29.2) | 948 (37.5) | 1840 (27.8) | 2260 (25.8)
Statistical Analysis 1: Comparison: BI 730357 25 mg Fast vs BI 730357 50 mg Fast vs BI 730357 100 mg Fast vs BI 730357 200 mg Fast; Dose proportionality for Cmax,ss of BI 730357 in plasma - fasted groups was assessed using a power model (regression model applied to log-transformed data); Test type: Other; Slope = 0.6005, 95% CI 2-sided [0.4534 to 0.7477], Standard Error of Mean 0.0722; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 730357 50 mg Fed vs BI 730357 200 mg Fed vs BI 730357 400 mg Fed; Dose proportionality for Cmax,ss of BI 730357 in plasma - fed groups was assessed using a power model (regression model applied to log-transformed data); Test type: Other; Slope = 0.5799, 95% CI 2-sided [0.4441 to 0.7156], Standard Error of Mean 0.0656; [other analysis details as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after last dose, up to 21 days (for 25, 50 and 100 mg dose groups) and up to 35 days (for 200 and 400 mg dose groups)
Description: Treated Set: This subject set included all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment. (One subject was orally administered mixed treatment of BI 730357 50 mg fast and placebo fast, thus evaluated twice in each respective treatment arm).
Arm/Group | Placebo Fast | Placebo Fed | BI 730357 25 mg Fast | BI 730357 50 mg Fast | BI 730357 50 mg Fed | BI 730357 100 mg Fast | BI 730357 200 mg Fast | BI 730357 200 mg Fed | BI 730357 400 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/9 | 0/10 | 0/8 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/9 | 0/10 | 0/8 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 8/12 | 5/9 | 7/9 | 6/10 | 7/8 | 4/9 | 8/9 | 4/9 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Fast (N=12) | Placebo Fed (N=9) | BI 730357 25 mg Fast (N=9) | BI 730357 50 mg Fast (N=10) | BI 730357 50 mg Fed (N=8) | BI 730357 100 mg Fast (N=9) | BI 730357 200 mg Fast (N=9) | BI 730357 200 mg Fed (N=9) | BI 730357 400 mg Fed (N=9)
Headache (Nervous system disorders) | 4 | 3 | 2 | 3 | 1 | 2 | 4 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT03279978/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT03279978/SAP_001.pdf